CLINICAL TRIAL: NCT05099406
Title: Brain and Pain (BaP): Understanding the Central Mechanisms of Pain to Improve Management of Patients With Refractory Chronic Pain
Brief Title: Home-based Transcranial Stimulation in the Treatment of Patients With Refractory Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government); Health Research Institute of Santiago de Compostela - IDIS (Recruitment support) (Unknown); Fundación Biomédica Galicia Sur (Recruitment support) (Unknown)
Responsible Party: Principal Investigator, María Teresa Carrillo de la Peña, Titular university professor (PhD), University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-PN133; 2021-000804-39 (EudraCT Number)
Record Dates: First submitted 2021-08-30; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Chronic Pain
Keywords: Transcranial electrical stimulation; Fibromyalgia; Arthritis; Arthrosis; Low back pain; Migraine headaches; Anxiety disorders; Depression; Chronic fatigue; Sleep disorders; Pain assessment; EEG
MeSH Terms: conditions — Chronic Pain; Fibromyalgia; Arthritis; Osteoarthritis; Low Back Pain; Migraine Disorders; Anxiety Disorders; Depression; Sleep Wake Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three treatment groups (40% active tDCS; 40% Active tACS; 20% Sham). Patients receiving sham stimulation will act as the control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Portable devices for applying the transcranial electrical stimulation are equipped with a software which allows a double-blinded procedure. The same computer program is in charge of randomly allocating patients to one of the three treatment groups. Thus, nor the researchers neither the participants will know what kind of stimulation is receiving each of them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Transcranial direct current stimulation (tDCS) (Active Comparator): Fifteen stimulation sessions applied with a daily frequency during an uninterrupted period of time which comprises just over two weeks. Current intensity of 2mA is applied during 20 minutes at the left M1, with anodal electrode placed in C3 and cathodal in FP2, following the International 10-20 EEG System. Ramp-up and ramp-down comprises 15 seconds at the beginning and end of the stimulation period.
  Interventions: Device: Transcranial electrical stimulation
- Transcranial alternant current stimulation (tACS) (Active Comparator): Fifteen stimulation sessions applied with a daily frequency during an uninterrupted period of time which comprises just over two weeks. Two electrodes will be placed at F3 and F4 and connected together for 10-Hz tACS (or the frequency which shows best sensitivity or specificity), and one electrode at Pz will be the return electrode. This setting is used to stimulate the somatosensory cortical region. Stimulation will last for 20 minutes, with a ramp-up and ramp-down of 15 seconds at the beginning and end of the session.
  Interventions: Device: Transcranial electrical stimulation
- Sham stimulation (Placebo Comparator): The electrode montage will be either the tDCS (for half of the participants) or the tACS montage (for the other half), and we will just apply the current at the ramps terms, but no current in the interval between the ramps which practically comprises the whole session. As for the two other group, fifteen sham stimulation sessions will be daily scheduled in a non-interrupted period of two weeks.
  Interventions: Device: Transcranial electrical stimulation

INTERVENTIONS:
Device: Transcranial electrical stimulation — By applying a low current over the cortex through the scalp, this technique can excite or inhibit the neural activity, thus modulating brain processes like pain perception and inducing relatively sustained changes in cortical excitability and neuroplasticity.
  Home-based transcranial electrical stimulation device consists of a custom headgear with fixed electrode sites and built-in cabling made for a simplistic setup for tDCS/tACS stimulation. Systems are equipped with strict dose control feature that provide reliable control over the intensity and timing of stimulation, turning these devices into a feasible and safe clinical alternative. The equipment is specifically designed for easy and simplistic self-setup and allows the researchers to remotely check the position of electrodes and also monitor the stimulation session.
  Other Names: Transcranial direct current stimulation; Transcranial alternant current stimulation

SUMMARY:
Refractory chronic pain represents a serious and limiting health condition which does not respond to standard pharmacological therapy. Thus, it emerges the necessity of new techniques to treat these group of diseases, such as the transcranial electrical stimulation (tES). This procedure induces a low-intensity electrical current through the scalp to modify the excitability of brain cells, thus facilitating changes in neural networks which may be dysfunctional in some chronic pain patients.

The main objective of this research is to test the efficacy of two tES techniques, differentiated by applying direct or alternant electrical current, to reduce the pain intensity and to increase pain thresholds of these patients. Besides, intervention is implemented at home for patients themselves thanks to a portable and convenient stimulator device, after one training session provided by technicians. Researches can supervise the compliance of the treatment remotely, as the stimulator has a permanent connection with their computers. A home-based approach means a more comfortable and accessible treatment alternative for patients, since they do not have to attend to clinics everyday to receive the stimulation; the advantages become even more relevant in the pandemic context, since the risk of being infected is radically minimized.

Despite the main purpose is to test the efficacy of tES to improve the pain suffered by patients, many other areas are considered as secondary end points for being intrinsically linked or affected by the disease, such as the interference in daily tasks provoked by pain, mood disorders (depression/anxiety), fatigue, life quality, physical functioning and sleep quality; these last two variables are measured with actigraph wristwatches, apart from specific questionnaires. Lastly, endogenous modulatory pain mechanisms are examined through sensory tests, namely Conditioned Pain Modulation and Temporal Summation of pain.

DETAILED DESCRIPTION:
This work aims to provide answers to the refractory chronic pain challenge. Pain is defined as refractory when multiple evidence-based biomedical therapies have failed to reach treatment goals that may include adequate pain reduction and/or improvement in daily functioning, even after appropriately assessing and addressing those psychosocial factors that could influence pain outcomes. In this sense, on the one hand, the study focus on detecting central biomarkers of pain modulation and processing which will contribute to improving knowledge of the mechanisms of pain chronification and the diagnosis procedure. On the other hand, given the low efficacy of pharmacological or non-pharmacological therapies for the patients studied, the efficacy of new therapeutic alternatives (tES) is explored. In short, the project will allow the transfer of knowledge to clinical practice in several aspects, such as diagnosis or treatment.

Therefore, the research aims to test the role of defective central pain modulation/processing as explanatory mechanisms for chronic pain. A second main objective is to test the efficacy of transcranial electric stimulation (tES) to modify dysfunction of central mechanism of pain, and to improve symptoms and quality of life in refractory chronic pain patients.

To achieve this, the investigators will select valid and reliable instruments to assess pain and comorbid symptoms in chronic pain patients and the most sensitive outcome measures to assess tES treatment efficacy. Sensory testing paradigms, namely Conditioned Pain Modulation, Temporal Summation of Second Pain and pain-related evoked potentials using electroencephalographic recordings, will act as biomarkers which are proposed to correlate with the severity of the chronic pain disease or some of their symptoms, and also as predictors of the treatment outcome.

Total sample includes 120 patients with refractory pharmaco-resistant pain, attended at the Pain Units of two Public Galician Hospitals (36 male, 84 female).

The study is expected to contribute to detection and preventive measures of future pain, and diagnosis of chronic pain disorders, improving prognosis and development of feasible patient-centered interventions, providing new directions for future research on pain.

ELIGIBILITY:
Inclusion Criteria:

* Suffering a chronic pain condition of non-cancer nature. Those patients who report chronic pain even after overcoming an oncological process are suitable to participate, but only if they have received the definitive medical discharge and have been free from radiotherapy/chemotherapy for at least twelve months.
* Adult subjects (18-65 years old).
* Subjects able to provide informed consent to participate in the study and to self-report pain.
* Existing chronic pain which reaches an intensity of at least 4 on a 0-10 Numeric Rating Scale (NRS) on average over the past 3 months prior to enrolment.
* Pain intensity of at least 5 on a 0-10 NRS over the week prior to enrolment.
* Diagnosis of pharmaco-resistance to analgesic drugs across the WHO ladder.
* Pharmacological regimen have kept stable for at least two months previous to the enrolment, and it must not suffer modifications during the whole research period.

Exclusion Criteria:

* Chronic pain derived from current cancer disease.
* Pregnant women or women in fertile age not having efficacious contraception during the whole period of the study.
* History of alcohol or drug abuse within the past 6 months as self-reported.
* Suffering from unstable medical conditions (e.g., uncontrolled diabetes, uncompensated cardiac issues, heart failure or chronic obstructive pulmonary disease).
* Intracranial ferromagnetic devices or implanted stimulator (basal ganglia stimulator, vagus nerve stimulation).
* Antecedents of, or active epilepsy.
* History of neurosurgery, psychiatric diseases other than anxiety or depression, traumatic brain injury with loss of consciousness, and/or cortical lesions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported pain intensity | Pre-treatment measure is the average of pain intensity of fifteen days previous to treatment; whereas the post-treatment measure is the average of fifteen days after treatment have finished
  Participants must evaluate the intensity of their pain using an online version of a Numerical Rating Scale of eleven points (0-10), so that the higher the score is, the worse the pain is.

SECONDARY OUTCOMES:
Global severity of chronic pain syndrome | Participants will complete MPI one or two days before the treatment onset, and one or two days after treatment ending.
  Composed index about the gravity of the chronic pain condition, taking into account several parameters as social and professional limitations due to pain, frequency and intensity of pain crisis, among others. The severity of chronic pain syndrome is assessed with global and subscales scores of Multidimensional Pain Inventory (MPI). Higher scores are indicative of worse health condition.
Pressure pain threshold | Pressure pain thresholds will be assessed in face-to-face laboratory sessions, which would take place one or two days before the treatment onset and one or two days after treatment ending.
  Pressure pain threshold is defined as the minimum force necessary to induce pain in the participant, measured using a manual algometer and operationalized in kPa.
Heat pain threshold | Heat pain thresholds will be assessed in face-to-face laboratory sessions, which would take place one or two days before the treatment onset and one or two days after treatment ending.
  Heat pain threshold is stablished as the temperature, measured in degrees Celsius, at which participant starts to feel pain, using a thermal stimulator.
Interference in daily living caused by pain | Pain interference will be assessed in face-to-face laboratory sessions, which would take place one or two days before the treatment onset and one or two days after treatment ending.
  Subscales of Multidimensional Pain Inventory (MPI) are used to evaluate whether patients usually leave undone or are not capable to do some daily activities and tasks due to the pain they suffer from. The test consists of a numerical rating scale of seven points (0-6), so that the higher the score is, the more pronounced is the interference due to pain.
Life quality | Life quality will be assessed one or two days before the treatment onset and one or two days after treatment ending.
  General health status considering physical, emotional and social functionality, as well as physical and mental health. Life quality is measured using the Short Form-36 Health Survey (SF-36). Higher scores are indicative of better health condition.
Physical condition and functioning | Estimations about daily energy expenditure, based on sedentary and activity bouts are recorded with wristband actigraphs which participants must wear during the whole research period.
  Involvement and time-spent in physical activities or exercises.
Sleep quality and disturbances | Participants will complete PQSI at two time-points, this is, one or two days before the treatment onset and one or two days after treatment ending.
  Sleep habits of participants and the degree in which they perceive that sleep as restorative. Sleep quality is measured using the Pittsburgh Sleep Quality Index (PSQI), a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Higher scores are indicative of poorer sleep quality.
Sleep quality and disturbances | Wristband actigraph are given to patients fifteen days before the treatment onset, so sleep habits are monitorized since that moment, until fifteen days after treatment have finished
  Sleep habits of participants, as total sleep time. This sleep parameter is measured using the data recorded for wristband actigraphs which participants must wear during the whole research period.
Pain unpleasantness | Pre-treatment measure is the average of pain unpleasantness obtained from fifteen daily assessments previous to treatment; whereas the post-treatment measure is the average obtained from the fifteen days after treatment have finished
  Affective component of pain, which refers to the discomfort or distress which pain provokes in patients. Participants must evaluate the discomfort produced by pain using an online version of a Numerical Rating Scale of eleven points (0-10), so that the higher the score is, the more stressful the pain is.
Mood disorders | Participants will complete HADS at two time-points, this is, one or two days before the treatment onset and one or two days after treatment ending.
  Depressive and anxiety symptomatology which can concur with chronic pain conditions. Mood alterations are measured using the Hospital Anxiety and Depression Scale (HADS). Higher scores are indicative of a worse mood state.
Anxiety | Pre-treatment measure is the average of anxiety levels obtained from fifteen daily assessments previous to treatment; whereas the post-treatment measure is the average obtained from the fifteen days after treatment have finished
  General anxiety level are evaluated with a daily frequency using an online version of a Numerical Rating Scale of eleven points (0-10), so that the higher the score is, the higher the anxiety level is.
Fatigue | Fatigue is registered with a daily frequency since the fifteen days before the treatment onset, until fifteen days after treatment ending. Participants will complete the MFIS at two time-points, this is, one or two days before and after treatment.
  Tiredness which may result in difficulties to perform physical or psychological tasks. Fatigue and its consequences are measured using the Modified Impact Fatigue Scale (MFIS). Numerical Rating Scales of eleven points (0-10) are also used to assess daily fatigue levels. In both cases, higher scores are indicative of a greater fatigue.
Caregiver burden | Caregivers are invited to a face-to-face interview with researchers one or two days before the treatment onset and one or two days after treatment ending.
  Stress levels which are subjected the caregivers of chronic pain patients are evaluated through the Zarit Burden Interview (ZBI) to assess if tES treatment means a reduction in burden derived from caring tasks. Higher scores are indicative of a more pronounced caregiver burden.
Global satisfaction with treatment and self-perceived improvement | Participants will evaluate their satisfaction with treatment a few days after it had finished.
  Patients are asked to rate their satisfaction with the tES treatment and whether they believe it has helped to improve their health status, using an ad-hoc designed questionnaire.

OTHER OUTCOMES:
Endogenous pain inhibition response | CPM procedure will be performed at two time-points, this is, one or two days before and after treatment, in order to assess if tES treatment is capable of restoring any dysfunction in this inhibitory pain network.
  Inhibitory pain system will be assessed through the Conditioned Pain Modulation (CPM) paradigm, which consists of the reduction of the pain provoked by a given noxious stimulus (i.e., test stimulus) when another painful stimulus (i.e., conditioning stimulus) is applied to a remote area (i.e., pain inhibits pain). Tentatively, we will use the cold water immersion of the non-dominant hand as conditioning stimuli; whereas the test stimuli will be the pressure pain thresholds using a digital handhold algometer, which puts progressively heavier pressure over the lateral area of dominant forearm. Differences in pressure pain threshold between the standard condition and when the CS is applied is assumed as an index of pain inhibitory response. Negative values are indicative of a greater pain inhibitory response.
Endogenous pain facilitation response | TSSP procedure will be performed at two time-points, this is, one or two days before and after treatment, in order to assess if tES treatment is capable of restoring any dysfunction in this facilitatory pain network.
  Amplifier pain system will be assessed through the Temporal Summation of Second Pain (TSSP) paradigm, which consists of the augmentation of subjective pain sensations due to the application of repeated noxious stimuli over the same corporal area, even when those stimuli are equal in terms of intensity and duration. Positive values are indicative of a greater pain facilitation score.
Electrical brain activity over diverse conditions | EEG will be registered at two time-points, this is, one or two days before and one or two days after treatment.
  Using the electroencephalography, we will capture the brain default mode network of chronic pain patients. Besides, we will register the evoked potentials elicited by diverse types of noxious heat-stimuli, as they may be reflecting how nociceptive signals are processed by brain. We purport to make a time-frequency and connectivity analysis of the EEG paying special attention to those key frequency bands involved in nociceptive perception, such as theta, alpha and gamma bands.

CONTACTS AND LOCATIONS:
Overall Officials: María Teresa Carrillo de la Peña, Principal Investigator — University of Santiago de Compostela
Locations (1):
- University of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn S, Prim JH, Alexander ML, McCulloch KL, Frohlich F. Identifying and Engaging Neuronal Oscillations by Transcranial Alternating Current Stimulation in Patients With Chronic Low Back Pain: A Randomized, Crossover, Double-Blind, Sham-Controlled Pilot Study. J Pain. 2019 Mar;20(3):277.e1-277.e11. doi: 10.1016/j.jpain.2018.09.004. Epub 2018 Sep 27. PMID 30268803
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Background] Arendt-Nielsen L, Nie H, Laursen MB, Laursen BS, Madeleine P, Simonsen OH, Graven-Nielsen T. Sensitization in patients with painful knee osteoarthritis. Pain. 2010 Jun;149(3):573-581. doi: 10.1016/j.pain.2010.04.003. Epub 2010 Apr 24. PMID 20418016
- [Background] Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333. doi: 10.1016/j.ejpain.2005.06.009. Epub 2005 Aug 10. PMID 16095934
- [Background] Bushnell MC, Ceko M, Low LA. Cognitive and emotional control of pain and its disruption in chronic pain. Nat Rev Neurosci. 2013 Jul;14(7):502-11. doi: 10.1038/nrn3516. Epub 2013 May 30. PMID 23719569
- [Background] Choe MK, Lim M, Kim JS, Lee DS, Chung CK. Disrupted Resting State Network of Fibromyalgia in Theta frequency. Sci Rep. 2018 Feb 1;8(1):2064. doi: 10.1038/s41598-017-18999-z. PMID 29391478
- [Background] Davis KD, Flor H, Greely HT, Iannetti GD, Mackey S, Ploner M, Pustilnik A, Tracey I, Treede RD, Wager TD. Brain imaging tests for chronic pain: medical, legal and ethical issues and recommendations. Nat Rev Neurol. 2017 Oct;13(10):624-638. doi: 10.1038/nrneurol.2017.122. Epub 2017 Sep 8. PMID 28884750
- [Background] De Keyser R, van den Broeke EN, Courtin A, Dufour A, Mouraux A. Event-related brain potentials elicited by high-speed cooling of the skin: A robust and non-painful method to assess the spinothalamic system in humans. Clin Neurophysiol. 2018 May;129(5):1011-1019. doi: 10.1016/j.clinph.2018.02.123. Epub 2018 Mar 8. PMID 29567583
- [Background] de Tommaso M, Ricci K, Libro G, Vecchio E, Delussi M, Montemurno A, Lopalco G, Iannone F. Pain Processing and Vegetative Dysfunction in Fibromyalgia: A Study by Sympathetic Skin Response and Laser Evoked Potentials. Pain Res Treat. 2017;2017:9747148. doi: 10.1155/2017/9747148. Epub 2017 Sep 28. PMID 29093972
- [Background] Duenas M, Salazar A, Ojeda B, Fernandez-Palacin F, Mico JA, Torres LM, Failde I. A nationwide study of chronic pain prevalence in the general spanish population: identifying clinical subgroups through cluster analysis. Pain Med. 2015 Apr;16(4):811-22. doi: 10.1111/pme.12640. Epub 2014 Dec 19. PMID 25530229
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Fallon N, Chiu Y, Nurmikko T, Stancak A. Altered theta oscillations in resting EEG of fibromyalgia syndrome patients. Eur J Pain. 2018 Jan;22(1):49-57. doi: 10.1002/ejp.1076. Epub 2017 Jul 31. PMID 28758313
- [Background] Fernandes C, Pidal-Miranda M, Samartin-Veiga N, Carrillo-de-la-Pena MT. Conditioned pain modulation as a biomarker of chronic pain: a systematic review of its concurrent validity. Pain. 2019 Dec;160(12):2679-2690. doi: 10.1097/j.pain.0000000000001664. PMID 31365469
- [Background] Frohlich F, Sellers KK, Cordle AL. Targeting the neurophysiology of cognitive systems with transcranial alternating current stimulation. Expert Rev Neurother. 2015 Feb;15(2):145-67. doi: 10.1586/14737175.2015.992782. Epub 2014 Dec 30. PMID 25547149
- [Background] Gonzalez-Villar AJ, Arias M, Carrillo-de-la-Pena MT. Brain Electrical Activity Associated With Visual Attention and Reactive Motor Inhibition in Patients With Fibromyalgia. Psychosom Med. 2019 May;81(4):380-388. doi: 10.1097/PSY.0000000000000677. PMID 31048636
- [Background] Jensen MP, Moore MR, Bockow TB, Ehde DM, Engel JM. Psychosocial factors and adjustment to chronic pain in persons with physical disabilities: a systematic review. Arch Phys Med Rehabil. 2011 Jan;92(1):146-60. doi: 10.1016/j.apmr.2010.09.021. PMID 21187217
- [Background] Hu L, Peng W, Valentini E, Zhang Z, Hu Y. Functional features of nociceptive-induced suppression of alpha band electroencephalographic oscillations. J Pain. 2013 Jan;14(1):89-99. doi: 10.1016/j.jpain.2012.10.008. PMID 23273836
- [Background] Keefe FJ, Rumble ME, Scipio CD, Giordano LA, Perri LM. Psychological aspects of persistent pain: current state of the science. J Pain. 2004 May;5(4):195-211. doi: 10.1016/j.jpain.2004.02.576. PMID 15162342
- [Background] Kosek E, Ordeberg G. Lack of pressure pain modulation by heterotopic noxious conditioning stimulation in patients with painful osteoarthritis before, but not following, surgical pain relief. Pain. 2000 Oct;88(1):69-78. doi: 10.1016/S0304-3959(00)00310-9. PMID 11098101
- [Background] Langley PC, Ruiz-Iban MA, Molina JT, De Andres J, Castellon JR. The prevalence, correlates and treatment of pain in Spain. J Med Econ. 2011;14(3):367-80. doi: 10.3111/13696998.2011.583303. Epub 2011 May 17. PMID 21574899
- [Background] Lefaucheur JP. A comprehensive database of published tDCS clinical trials (2005-2016). Neurophysiol Clin. 2016 Dec;46(6):319-398. doi: 10.1016/j.neucli.2016.10.002. Epub 2016 Nov 17. PMID 27865707
- [Background] Lewis GN, Rice DA, McNair PJ. Conditioned pain modulation in populations with chronic pain: a systematic review and meta-analysis. J Pain. 2012 Oct;13(10):936-44. doi: 10.1016/j.jpain.2012.07.005. Epub 2012 Sep 13. PMID 22981090
- [Background] Alappat JJ. Motor cortex stimulation for chronic pain: systematic review and meta-analysis of the literature. Neurology. 2009 Feb 10;72(6):577; author reply 577. doi: 10.1212/01.wnl.0000344169.51931.e5. No abstract available. PMID 19204274
- [Background] Maarrawi J, Peyron R, Mertens P, Costes N, Magnin M, Sindou M, Laurent B, Garcia-Larrea L. Motor cortex stimulation for pain control induces changes in the endogenous opioid system. Neurology. 2007 Aug 28;69(9):827-34. doi: 10.1212/01.wnl.0000269783.86997.37. PMID 17724284
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] O'Brien AT, Deitos A, Trinanes Pego Y, Fregni F, Carrillo-de-la-Pena MT. Defective Endogenous Pain Modulation in Fibromyalgia: A Meta-Analysis of Temporal Summation and Conditioned Pain Modulation Paradigms. J Pain. 2018 Aug;19(8):819-836. doi: 10.1016/j.jpain.2018.01.010. Epub 2018 Feb 15. PMID 29454976
- [Background] Peng W, Tang D. Pain Related Cortical Oscillations: Methodological Advances and Potential Applications. Front Comput Neurosci. 2016 Feb 4;10:9. doi: 10.3389/fncom.2016.00009. eCollection 2016. PMID 26869915
- [Background] Petersen KK, Arendt-Nielsen L, Simonsen O, Wilder-Smith O, Laursen MB. Presurgical assessment of temporal summation of pain predicts the development of chronic postoperative pain 12 months after total knee replacement. Pain. 2015 Jan;156(1):55-61. doi: 10.1016/j.pain.0000000000000022. PMID 25599301
- [Background] Ploner M, Sorg C, Gross J. Brain Rhythms of Pain. Trends Cogn Sci. 2017 Feb;21(2):100-110. doi: 10.1016/j.tics.2016.12.001. Epub 2016 Dec 23. PMID 28025007
- [Background] Potvin S, Marchand S. Pain facilitation and pain inhibition during conditioned pain modulation in fibromyalgia and in healthy controls. Pain. 2016 Aug;157(8):1704-1710. doi: 10.1097/j.pain.0000000000000573. PMID 27045524
- [Background] Staud R, Vierck CJ, Cannon RL, Mauderli AP, Price DD. Abnormal sensitization and temporal summation of second pain (wind-up) in patients with fibromyalgia syndrome. Pain. 2001 Mar;91(1-2):165-75. doi: 10.1016/s0304-3959(00)00432-2. PMID 11240089
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. A classification of chronic pain for ICD-11. Pain. 2015 Jun;156(6):1003-1007. doi: 10.1097/j.pain.0000000000000160. No abstract available. PMID 25844555
- [Background] Woods AJ, Antal A, Bikson M, Boggio PS, Brunoni AR, Celnik P, Cohen LG, Fregni F, Herrmann CS, Kappenman ES, Knotkova H, Liebetanz D, Miniussi C, Miranda PC, Paulus W, Priori A, Reato D, Stagg C, Wenderoth N, Nitsche MA. A technical guide to tDCS, and related non-invasive brain stimulation tools. Clin Neurophysiol. 2016 Feb;127(2):1031-1048. doi: 10.1016/j.clinph.2015.11.012. Epub 2015 Nov 22. PMID 26652115
- [Background] Zortea M, Ramalho L, Alves RL, Alves CFDS, Braulio G, Torres ILDS, Fregni F, Caumo W. Transcranial Direct Current Stimulation to Improve the Dysfunction of Descending Pain Modulatory System Related to Opioids in Chronic Non-cancer Pain: An Integrative Review of Neurobiology and Meta-Analysis. Front Neurosci. 2019 Nov 18;13:1218. doi: 10.3389/fnins.2019.01218. eCollection 2019. PMID 31803005
- [Derived] Gil-Ugidos A, Alcantara-Espinosa J, Rubal-Otero L, Mayo-Moldes M, Samartin-Veiga N, Carrillo-de-la-Pena MT. Transcranial electrical stimulation (tES) in chronic pain patients: Effects on daily-reported symptoms. Anaesth Crit Care Pain Med. 2026 Jan;45(1):101613. doi: 10.1016/j.accpm.2025.101613. Epub 2025 Sep 25. PMID 41015289
- [Derived] Fernandez A, Rubal-Otero L, Gil-Ugidos A, Pinal D, Gonzalez-Villar AJ, Carrillo-de-la-Pena MT. Distinct resting state neural activity in chronic pain patients who respond to transcranial electric stimulation for pain relief. Front Hum Neurosci. 2025 Jul 15;19:1546414. doi: 10.3389/fnhum.2025.1546414. eCollection 2025. PMID 40735279

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT05099406/Prot_SAP_000.pdf